CLINICAL TRIAL: NCT03271320
Title: Evaluation of Aesthetic Impact in Patients With Systemic Sclerosis
Acronym: SCLERO-ESTHET
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_63; 2016-A00735-46 (Other: ID-RCB number)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systemic sclerosis: patients with systemic sclerosis
  Interventions: Other: appearance scales
- control: Healthy subjects
  Interventions: Other: appearance scales

INTERVENTIONS:
Other: appearance scales — appearance scales : AVS; ASWAP; DAS 59

SUMMARY:
The primary objective is to assess the burden of aesthetic complication in systemic sclerosis. Systemic sclerosis is associated with changes in skin aspect which can impact the appearance. Aesthetic burden will be assessed through several scales and compared to a control group of health subjects.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis according to ACR-EULAR 2013

Exclusion Criteria:

* non French native
* aesthetic sequel from other conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: systemic sclerosis patients
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Visual scale for aesthetic burden | Baseline
  Visual scale for aesthetic burden from 0 to 10

SECONDARY OUTCOMES:
Satisfaction with Appearance Scale (SWAP) | Baseline
  The SWAP measures body image dissatisfaction in persons with visible disfigurement
Derriford Appearance Scale-59 (DAS) | Baseline
  The Derriford Appearance Scales measure the spectrum of psychological distress and dysfunction that is characteristic of disfigurements, deformities and aesthetic problems of appearance.
Multidimensional Body self Relations Questionnaire (MBSRQ) | Baseline
  The Multidimensional Body-Self Relations Questionnaire (MBSRQ) is a 69-item self-report inventory for the assessment of self-attitudinal aspects of the body-image construct.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Claude Huriez, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farhat MM, Guerreschi P, Morell-Dubois S, Deken V, Labreuche J, Sanges S, Sobanski V, Hachulla E, Cottencin O, Launay D. Perception of aesthetic impairment in patients with systemic sclerosis determined using a semi-quantitative scale and its association with disease characteristics. J Scleroderma Relat Disord. 2024 Jun;9(2):124-133. doi: 10.1177/23971983241231620. Epub 2024 Feb 27. PMID 38910601